CLINICAL TRIAL: NCT02494115
Title: Comfort Subcutaneous Drainage: a Descriptive Study Among Palliative Care Cancer Patients Presenting Severe Refractory Lower Limbs Lymphedema
Brief Title: Comfort Subcutaneous Drainage: a Descriptive Study Among Palliative Phase Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-PP12
Record Dates: First submitted 2015-06-26; First posted 2015-07-10 (Estimated); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Lymphedema
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- subcutaneous drainage (Experimental): This local treatment consists in inserting in lower limbs several catheters draining into enclosed bags in order to evacuate lymph fluid and to lower local pressure.
  Interventions: Procedure: subcutaneous drainage

INTERVENTIONS:
Procedure: subcutaneous drainage

SUMMARY:
Physical embarrassment, pain and psychological impact linked to the body image distortion are often associated to these lymphedemas. Investigators decided to study new therapeutic method because of major discomfort due to these oedemas and doctors' difficulty to manage them.

Subcutaneous drainage also called lymphocentesis seems to be an interesting technique. This local treatment consists in inserting in lower limbs several catheters draining into enclosed bags in order to evacuate lymph fluid and to lower local pressure.

Very few studies have been published concerning this technique and are presenting only a small number of cases. They cannot allow clear conclusions of this technique's efficiency but show encouraging results.

Investigators want to collect more data on this technique using a larger number of subjects in order to evaluate subcutaneous drainage effects on the comfort of palliative care cancer patients presenting lower limbs lymphedema. Investigators will consider as lymphedema, oedemas with no renal or cardiovascular identified cause and excluding anasarca.

DETAILED DESCRIPTION:
Lower limbs lymphedemas are often reported in advanced palliative phase cancer patients. These oedemas have multiple causes and are complicated to be taken care of. Actual available treatments such as physiotherapist massage and compression stockings, are often lacking efficiency and are not adapted for these patients.

Physical embarrassment, pain and psychological impact linked to the body image distortion are often associated to these lymphedemas. Investigators decided to study new therapeutic method because of major discomfort due to these oedemas and doctors' difficulty to manage them.

Subcutaneous drainage also called lymphocentesis seems to be an interesting technique. This local treatment consists in inserting in lower limbs several catheters draining into enclosed bags in order to evacuate lymph fluid and to lower local pressure.

Very few studies have been published concerning this technique and are presenting only a small number of cases. They cannot allow clear conclusions of this technique's efficiency but show encouraging results.

Investigators want to collect more data on this technique using a larger number of subjects in order to evaluate subcutaneous drainage effects on the comfort of palliative care cancer patients presenting lower limbs lymphedema. Investigators will consider as lymphedema, oedemas with no renal or cardiovascular identified cause and excluding anasarca.

This study should be completed by a comparative randomized study to increase the evidence level if it shows a technical interest for drainage.

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients
* Palliative care patients according to the SFAP (French Palliative care society) definition
* Patient taken care of in one of the palliative care structures implied in this project (palliative care unit, palliative care field team, hospital at home, palliative care day hospital)
* Patients presenting lower limb lymphedema resistant to traditional treatments or for whom these treatments are not adapted
* Lymphedema being a source of discomfort for the patient asking for relief
* Patient wishing a new treatment for lymphedema
* Patients with full cognitive capacities evaluated by the practitioner in charge of him
* Patients available during the study

Exclusion Criteria:

* Lost-of-sight or transferred to another hospital subjects
* Subjects wishing to end their participation before study ending

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-01-06 (Actual); Primary Completion 2018-09-15 (Actual); Study Completion 2018-09-15 (Actual)

PRIMARY OUTCOMES:
evolution of the patient's discomfort due to his oedemas | on the 3rd day after lymphcentesis
  It will be measured with a numeric scale from 0 no discomfort to 10 maximal discomfort.

CONTACTS AND LOCATIONS:
Overall Officials: Flora TREMELLAT, MD, Principal Investigator — tremellat.f@chu-nice.fr
Locations (3):
- France (3):
  - CAL, Nice, Alpes-maritimes
  - Centre Hospitalier, Avignon
  - Centre Hospitalier Universitaire de Nice, Nice